CLINICAL TRIAL: NCT00642174
Title: A Pharmacodynamic Comparison of Prasugrel (LY640315) Versus High Dose Clopidogrel in Subjects With Type 2 Diabetes Mellitus and Coronary Artery Disease.
Brief Title: Third Optimizing Anti-Platelet Therapy in Diabetes MellitUS (OPTIMUS-3)
Acronym: OPTIMUS-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11241; H7T-MC-TACA (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-03-21; First posted 2008-03-24 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): Oral prasugrel 60-mg loading dose, followed by 6 to 9 days of prasugrel 10-mg/day tablet maintenance dose.
  Interventions: Drug: prasugrel
- Clopidogrel (Active Comparator): Oral clopidogrel 600-mg loading dose, followed by 6 to 9 days of clopidogrel 150-mg/day tablet maintenance dose.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: prasugrel — Oral prasugrel 60-mg loading dose, followed by 6-9 days of oral prasugrel 10-mg/day tablet maintenance dose.
  Other Names: LY640315; Effient; Efient
  Arms: Prasugrel
Drug: Clopidogrel — Oral clopidogrel 600-mg loading dose, followed by 6-9 days of oral clopidogrel 150-mg/day tablet maintenance dose.
  Arms: Clopidogrel

SUMMARY:
This trial is designed as a phase 2 randomized, double-blind double dummy, active comparator controlled, two-period two-arm crossover study to enroll 40 patients across multiple centers. The study will compare platelet function following a prasugrel loading dose and 1 week of prasugrel maintenance therapy with high-dose clopidogrel loading dose and 1 week of high-dose clopidogrel maintenance therapy in patients with drug treated type 2 diabetes mellitus who have coronary artery disease. Various assays of platelet function will be used in this study. Platelet function will be studied using the following assays: Accumetrics VerifyNowTM P2Y12, Light Transmittance Aggregometry (LTA), Vasodilator-associated stimulated phosphoprotein (VASP), and Thromboelastography (TEG)-platelet mapping.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus and on oral or parenteral hypoglycemic therapy for at least 1 month.
* History of Coronary Artery Disease with or without other types of vascular disease (such as peripheral vascular disease).
* Taking Aspirin 75-325 mg/day for at least 1 week prior to randomization.
* Between the ages of 18-74 years old.
* If a woman of child bearing age, must not be pregnant and must agree to use reliable method of birth control during the duration of the study.

Exclusion Criteria:

* Thienopyridine therapy within 30 days or have a defined need for thienopyridine treatment.
* Coronary Artery Bypass Graft (CABG) or Percutaneous Coronary Intervention (PCI) with no stent placed within 30 days.
* Planned coronary revascularization
* Hemoglobin A1c (HbA1c) > or equal to 10 mg/dL within the last 3 months.
* Received fibrolytic therapy <24 hours prior to randomization.
* Received non-fibrin-specific fibrinolytic therapy <48 hours prior to randomization.
* At risk of bleeding.
* History of ischemic stroke, transient ischemic attack (TIA), intercranial neoplasm, arteriovenous malformation, or aneurysm.
* Body weight <60 kilograms (kg).
* International Normalized Ratio (INR) >1.5, platelet count <100,000/mm3, or anemia (hemoglobin <10 gm/dL) within 1 week of study entry.
* Are receiving or will receive oral anticoagulation or antiplatelet treatment therapy.
* Are being treated with daily non-steroidal anti-inflammatory drugs (NSAIDS).
* Are pregnant, breast-feeding or plan to become pregnant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am-5pm Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Angiolillo DJ, Badimon JJ, Saucedo JF, Frelinger AL, Michelson AD, Jakubowski JA, Zhu B, Ojeh CK, Baker BA, Effron MB. A pharmacodynamic comparison of prasugrel vs. high-dose clopidogrel in patients with type 2 diabetes mellitus and coronary artery disease: results of the Optimizing anti-Platelet Therapy In diabetes MellitUS (OPTIMUS)-3 Trial. Eur Heart J. 2011 Apr;32(7):838-46. doi: 10.1093/eurheartj/ehq494. Epub 2011 Jan 20. PMID 21252171
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel Then Clopidogrel: Prasugrel: Oral prasugrel 60-mg loading dose, followed by 6 to 9 days of prasugrel 10-mg/day tablet maintenance dose. Clopidogrel: Oral clopidogrel 600-mg loading dose, followed by 6 to 9 days of clopidogrel 150-mg/day tablet maintenance dose.
- Clopidogrel Then Prasugrel: Clopidogrel: Oral clopidogrel 600-mg loading dose, followed by 6 to 9 days of clopidogrel 150-mg/day tablet maintenance dose. Prasugrel: Oral prasugrel 60-mg loading dose, followed by 6 to 9 days of prasugrel 10-mg/day tablet maintenance dose.
Period: Period 1 - Initial Drug
Arm/Group | Prasugrel Then Clopidogrel | Clopidogrel Then Prasugrel
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1
Not completed — Entry Criteria Not Met | 0 | 1
Period: Period 2 - Crossover Drug
Arm/Group | Prasugrel Then Clopidogrel | Clopidogrel Then Prasugrel
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel Then Clopidogrel | Clopidogrel Then Prasugrel | Total
Number analyzed (Participants) | 18 | 17 | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.43) | 62.4 (8.14) | 61.3 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 14 | 10 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 | 7 | 15
  African | 3 | 4 | 7
  Hispanic | 4 | 4 | 8
  Native American | 0 | 1 | 1
  East Asian | 1 | 0 | 1
  West Asian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Platelet Aggregation (IPA) 4 Hours After Loading Dose Assessed by Accumetrics VerifyNow™ P2Y12 Assay
Description: The inhibition of platelet aggregation 4 hours after the loading dose was administered was assessed using the Accumetrics VerifyNow™ P2Y12 assay. Percentage inhibition, as reported by VerifyNow™ P2Y12, was calculated from P2Y12 Reaction Unit (PRU) (rate and extent of adenosine diphosphate [ADP]-stimulated platelet aggregation) and BASE (estimate of baseline platelet reactivity independent of P2Y12 receptor inhibition [reference values]: rate and extent of Thrombin Receptor-Activated Peptide-stimulated platelet aggregation) values as follows: Percentage (%) inhibition = (1-PRU/BASE) x 100.
Time Frame: 4 hours after loading dose
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for IPA at 4 hours, who met compliance criteria, and who had last dose of study drug prior to the blood draw for IPA.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent inhibition
Groups:
- Prasugrel: Prasugrel: Oral prasugrel 60-mg loading dose, followed by 6 to 9 days of prasugrel 10-mg/day tablet maintenance dose.
- Clopidogrel: Clopidogrel: Oral clopidogrel 600-mg loading dose, followed by 6 to 9 days of clopidogrel 150-mg/day tablet maintenance dose.
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 34 | 35
percent inhibition
  Baseline | 9.4 (10.23) [5.55 to 13.18] | 9.3 (11.46) [5.55 to 13.15]
  4 Hours After Loading Dose | 89.3 (9.40) [82.96 to 95.60] | 27.7 (23.82) [21.49 to 33.94]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Null hypothesis: there is no difference between prasugrel and clopidogrel in IPA assessed by Accumetrics VerifyNow™ P2Y12 4 hours after administration of loading dose. Assuming 90% power, 2-sided alpha of 0.05, and a 17.5% difference in IPA between treatment groups with a standard deviation of 20, a total of 15 completed subjects per sequence group (i.e., 15 subject who receive prasugrel first, then clopidogrel; and 15 subjects who receive clopidogrel first, then prasugrel) was determined; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for 4 Hours After Loading Dose; Linear mixed model with treatment, sequence and treatment by sequence (i.e. period) as fixed effects and subject as random effect; Least Squares Mean Difference (Net) = 61.6, 95% CI [53.83 to 69.31] — Least Squares Mean Difference = Prasugrel minus Clopidogrel

2. Secondary Outcome: Inhibition of Platelet Aggregation at 1- and 24-Hours After Loading Dose (LD) and 24-Hours After Last Maintenance Dose (LMD) Assessed by Accumetrics VerifyNow™ P2Y12 Assay
Description: Inhibition of platelet aggregation 1- and 24-hours after loading dose and 24-hours after last maintenance dose was administered was assessed using Accumetrics VerifyNow™ P2Y12 assay. Percentage inhibition, as reported by VerifyNow™ P2Y12, was calculated from PRU (rate and extent of ADP-stimulated platelet aggregation) and BASE (estimate of baseline platelet reactivity independent of P2Y12 receptor inhibition [reference values]: rate and extent of Thrombin Receptor-Activated Peptide-stimulated platelet aggregation) values as follows: Percentage (%) inhibition = (1-PRU/BASE) x 100.
Time Frame: 1 hour and 24 hours after the loading dose (LD) and 24 hours after the last maintenance dose (LMD)
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for IPA, who met compliance criteria, and who had last dose of study drug prior to the blood draw for IPA.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 34 | 35
percent inhibition
  1 Hour After Loading Dose | 49.9 [41.17 to 58.60] | 13.4 [4.92 to 21.89]
  24 Hours After Loading Dose | 87.1 [80.64 to 93.66] | 29.3 [22.87 to 35.68]
  24 Hours After Last Maintenance Dose | 61.8 [55.70 to 67.91] | 44.2 [38.05 to 50.26]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Null hypothesis: there was no difference between prasugrel and clopidogrel in IPA assessed by Accumetrics VerifyNow™ P2Y12 1 hour after administration of the loading dose; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 1 Hour After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; Linear mixed model with treatment, sequence and treatment by sequence (ie. period) as fixed effects and subject as random effect; Mean Difference (Net) = 36.5, 95% CI [27.43 to 45.52] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; Null hypothesis: there was no difference between prasugrel and clopidogrel in IPA assessed by Accumetrics VerifyNow™ P2Y12 24 hours after administration of the loading dose; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hour After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 57.9, 95% CI [49.56 to 66.19] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; Null hypothesis: there was no difference between prasugrel and clopidogrel in IPA assessed by Accumetrics VerifyNow™ P2Y12 24 hours post-Last Maintenance Dose (LMD); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hours After Last Maintenance Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 17.7, 95% CI [10.27 to 25.04] — Least Squares Mean Difference = Prasugrel minus Clopidogrel

3. Secondary Outcome: Maximum Platelet Aggregation (MPA) as Assessed by Light Transmittance Aggregometry (LTA)
Description: Mean platelet aggregation (MPA) to 5 and 20 µM adenosine diphosphate (ADP) was assessed by light transmittance aggregometry (LTA). Platelet aggregation was monitored for a total of 7 minutes after addition of ADP. Maximum platelet aggregation was the maximal aggregation value achieved during the 7-minute observation period following addition of agonists.
Time Frame: Baseline, 1 Hour, 4 Hours, and 24 Hours after loading dose, and 24 Hours after last maintenance dose
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for MPA, who met compliance criteria, and who had last dose of study drug prior to the blood draw for MPA.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent platelet aggregation
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 34 | 35
percent platelet aggregation
  Baseline (5 μM ADP) | 64.9 [61.62 to 68.14] | 65.7 [62.49 to 68.95]
  1 Hour After Loading Dose (5 μM ADP) | 33.7 [28.44 to 39.03] | 56.7 [51.69 to 61.77]
  4 Hours After Loading Dose (5 μM ADP) | 18.0 [13.41 to 22.51] | 44.6 [40.11 to 49.00]
  24 Hours After Loading Dose (5 μM ADP) | 22.3 [17.78 to 26.89] | 45.6 [41.20 to 50.06]
  24 Hours After Last Maintenance Dose (5 μM ADP) | 29.6 [25.20 to 34.08] | 38.3 [33.93 to 42.71]
  Baseline (20 μM ADP) | 77.1 [73.74 to 80.43] | 76.9 [73.54 to 80.17]
  1 Hour After Loading Dose (20 μM ADP) | 44.7 [38.54 to 50.77] | 69.8 [64.05 to 75.56]
  4 Hours After Loading Dose (20 μM ADP) | 22.4 [16.99 to 27.81] | 57.5 [52.16 to 62.75]
  24 Hours After Loading Dose (20 μM ADP) | 27.4 [22.23 to 32.67] | 58.4 [53.39 to 63.48]
  24 Hours After Last Maintenance Dose (20 μM ADP) | 38.3 [32.97 to 43.64] | 50.7 [45.42 to 55.97]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; The null hypothesis was that there was no difference between prasugrel and clopidogrel in MPA assessed by Light Transmittance Aggregometry (LTA); Test type: Superiority or Other; p = 0.5466, Mixed Models Analysis — P-value for Baseline (5 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.8, 95% CI [-3.66 to 1.97] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 1 After Post Loading Dose (5 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -23.0, 95% CI [-28.45 to -17.55] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 Hour After Loading Dose (5 uM ADP). A priori threshold for statisitical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -26.6, 95% CI [-31.18 to -22.02] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 4: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hour After Loading Dose (5 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -23.3, 95% CI [-27.42 to -19.17] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 5: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — P-value for 24 Hour After Last Maintenance Dose (5 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -8.7, 95% CI [-12.78 to -4.58] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 6: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8779, Mixed Models Analysis — P-value for Baseline (20 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 0.2, 95% CI [-2.80 to 3.26] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 7: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 1 Hour After Loading Dose (20 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -25.2, 95% CI [-32.43 to -17.87] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 8: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 Hour After Loading Dose (20 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -35.1, 95% CI [-40.32 to -29.78] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 9: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hour After Loading Dose (20 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -31.0, 95% CI [-36.32 to -25.66] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 10: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hour After Last Maintenance Dose (20 uM ADP). A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -12.4, 95% CI [-17.19 to -7.58] — Least Squares Mean Difference = Prasugrel minus Clopidogrel

4. Secondary Outcome: Platelet Reactivity Index (PRI)
Description: Data from the Vasodilator-associated stimulated phosphoprotein assay were reported as the platelet reactivity index (PRI) which was calculated from corrected mean fluorescence intensity (cMFI) following incubation of platelets with either prostaglandin E1 (PGE1) alone or PGE1 plus ADP: Platelet Reactivity Index (%) = [1-(cMFI PGEI+ADP/cMFI PGEI)] x 100. Lower PRI values indicate greater platelet P2Y12 inhibition.
Time Frame: Baseline, 1 Hour, 4 Hours, and 24 Hours after loading dose, and 24 Hours after last maintenance dose
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for Vasodilator-Associated Stimulated Phosphoprotein (VASP), who met compliance criteria, and who had last dose of study drug prior to the blood draw for inhibition of platelet function as assessed by VASP.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 34 | 35
percent inhibition
  Baseline | 83.5 [78.76 to 88.31] | 80.6 [75.92 to 85.31]
  1 Hour After Loading Dose | 40.0 [32.14 to 47.80] | 76.2 [68.48 to 83.88]
  4 Hours After Loading Dose | 14.5 [7.73 to 21.35] | 67.5 [60.79 to 74.19]
  24 Hours After Loading Dose | 15.7 [8.33 to 22.99] | 58.5 [51.30 to 65.61]
  24 Hours After Last Maintenance Dose | 27.4 [20.82 to 34.03] | 42.3 [35.72 to 48.93]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; The null hypothesis was that there was no difference between prasugrel and clopidogrel in Inhibition of Platelet Function as assessed by VASP; Test type: Superiority or Other; p = 0.3692, Mixed Models Analysis — P-value for Baseline. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 2.9, 95% CI [-3.60 to 9.44] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 1 Hour After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -36.2, 95% CI [-47.43 to -24.98] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 Hours After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -53.0, 95% CI [-61.89 to -44.02] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 4: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hours After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -42.8, 95% CI [-50.03 to -35.55] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 5: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis — P-value for 24 Hours After Last Maintenance Dose. A priori threshold for statistical significance was set to p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -14.9, 95% CI [-23.42 to -6.37] — Least Squares Mean Difference = Prasugrel minus Clopidogrel

5. Secondary Outcome: Inhibition of Platelet Function as Measured by Thromboelastography (TEG)-Platelet Mapping Maximum Amplitude - Adenosine Diphosphate
Description: Thromboelastography (TEG) platelet mapping (MP) maximum amplitude (MA) - Adenosine Diphosphate (ADP) millimeters (mm) at each time point. The TEG-MP MA measures strength of clot formation in whole blood. MA-ADP is the maximal amplitude resulting from fibrin and platelets not blocked by ADP-receptor inhibiting drugs. Fibrin strands in blood sample link a rotating sample cup with a stationary pin suspended by a torsion wire. The degree of platelet contribution to the MA through platelet-fibrin bonding directly influences the magnitude of pin movement and ultimately the amplitude of the tracing.
Time Frame: Baseline, 1 Hour, 4 Hours, and 24 Hours after loading dose, and 24 Hours after last maintenance dose
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for Inhibition of Platelet Function (IPF) as measured by Thromboelastography (TEG)-Platelet Mapping Maximum Amplitude - Adenosine Diphosphate (ADP), who met compliance criteria, and who had last dose of study drug prior to blood draw for IPF.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters (mm)
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 34 | 35
millimeters (mm)
  Baseline | 56.8 [52.37 to 61.21] | 58.1 [53.70 to 62.45]
  1 Hour After Loading Dose | 38.5 [33.42 to 43.63] | 54.8 [49.84 to 59.69]
  4 Hours After Loading Dose | 24.2 [18.80 to 29.6] | 48.1 [42.84 to 53.35]
  24 Hours After Loading Dose | 29.3 [24.56 to 34.01] | 49.2 [44.61 to 53.82]
  24 Hours After Last Maintenance Dose | 44.2 [38.77 to 49.62] | 46.8 [41.37 to 52.22]
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Null hypothesis: no difference between prasugrel and clopidogrel in Inhibition of Platelet Function as measured by Thromboelastography (TEG)-Platelet Mapping Maximum Amplitude - Adenosine Diphosphate (ADP); Test type: Superiority or Other; p = 0.5238, Mixed Models Analysis — P-value for Baseline. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.3, 95% CI [-5.35 to 2.78] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 2: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 1 Hour After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -16.2, 95% CI [-21.15 to -11.33] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 3: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 4 Hours After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -23.9, 95% CI [-29.67 to -18.11] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 4: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value for 24 Hours After Loading Dose. A priori threshold for statistical significance was set at p=0.05 level; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -19.9, 95% CI [-24.97 to -14.90] — Least Squares Mean Difference = Prasugrel minus Clopidogrel
Statistical Analysis 5: Comparison: Prasugrel vs Clopidogrel; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3725, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -2.6, 95% CI [-8.46 to 3.26] — Least Squares Mean Difference = Prasugrel minus Clopidogrel

ADVERSE EVENTS:
Arm/Group | Prasugrel | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 5/34 | 9/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=34) | Clopidogrel (N=35)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wart excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days